CLINICAL TRIAL: NCT00004649
Title: Study of the Natural History and Genotype-Phenotype Correlations of Hereditary Hemorrhagic Telangiectasia Patients
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Vermont (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11712; UVT-650
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: genetic diseases and dysmorphic syndromes; hematologic disorders; hereditary hemorrhagic telangiectasia; rare disease
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Collect data regarding the natural history of hereditary hemorrhagic telangiectasia (HHT).

II. Establish genotype-phenotype correlations in HHT. III. Create a database of information for researchers throughout the world.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients complete a self-administered natural history questionnaire in a multiple choice format. Questionnaire is completed by a population consisting of males and females of all ages and ethnic backgrounds.

Data are collected and made available to all researchers.

ELIGIBILITY:
* Diagnosed hereditary hemorrhagic telangiectasia (Osler-Rendu-Weber disease) with recurrent epistaxis, telangiectases, and visceral vascular anomalies

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-05

CONTACTS AND LOCATIONS:
Overall Officials: Alan Guttmacher, Study Chair — University of Vermont